CLINICAL TRIAL: NCT05752227
Title: Difference In Strain Ratio Ultrasound Elastography Between Benign And Malignant Peripheral Parenchymal Lung Lesions.
Brief Title: Difference Strain Ratio Ultrasound Elastography Between Benign and Malignant Peripheral Lung Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: 0201692
Record Dates: First submitted 2022-12-23; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-11

CONDITIONS: Peripheral Lung Lesions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- benign lung lesions: Patient who were diagnosed with peripheral lung lesions including consolidation, atelectasis, or cavitation
  Interventions: Procedure: Transthoracic biopsy; Radiation: CT chest
- malignant lung lesions: patients diagnosed with malignant lung lesions
  Interventions: Procedure: Transthoracic biopsy; Radiation: CT chest

INTERVENTIONS:
Procedure: Transthoracic biopsy — Us guided transthoracic biopsy
Radiation: CT chest — Computed tomography

SUMMARY:
Diagnostic accuracy study to investigate the sensitivity and specificity of sonographic elastography using strain ratio to differentiate between benign and malignant peripheral lesions in comparison to biopsy, clinically, or radiologically.

DETAILED DESCRIPTION:
This is a diagnostic accuracy study with comparison to gold standard tests e.g., chest computed tomography, transthoracic biopsy, or microbiological analysis. All patients included in this study will give informed consent according to the guidelines of ethics committee, Alexandria Faculty of Medicine. (http://www.med.alexu.edu.eg/wp-content/uploads/2012/04/Checklist-FINAL- 20141.pdf-)

ELIGIBILITY:
Inclusion Criteria:

* 1) Adult patients above age of 18 years old. 2) Patients with peripheral lung lesion.

Exclusion Criteria:

1. Pure pleural lesions.
2. Clinical instability to reach the final diagnosis.
3. Inaccessibility by ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Above age of 18 yrs old
Study Population: Patients are all above age of 18 yrs old without gender discrimination
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Cut off value strain ratio | 6-9 months
  To differentiate between benign and malignant lung lesions using strain ratio

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed F Abouelnour, Masters, Principal Investigator — Alexandrian University
Locations (1):
- Ahmed Farag Abouelnour, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and full methodology of our study to be shared
Supporting Information: Study Protocol, SAP
Time Frame: will be available within 6 months for 1 year
Access Criteria: abouelnourahmed@gmail.com

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT05752227/Prot_SAP_000.pdf